CLINICAL TRIAL: NCT06247228
Title: A Co-created Digital Intervention to Reduce Home-office Workers' Sedentary Behaviour: Protocol for the Click2Move Programme, a Cluster Randomised Controlled Trial
Brief Title: Click2Move Intervention to Reduce Home-office Workers' Sedentary Behaviour.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vic - Central University of Catalonia (Other)
Collaborators: National Institute for Public Health and the Environment (RIVM) (Other Government); Technological University of the Shannon, Athlone, Ireland (Unknown); University of Ljubljana (Other)
Responsible Party: Principal Investigator, Judit Bort, Principal Investigator, University of Vic - Central University of Catalonia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C2M278/2023
Record Dates: First submitted 2024-01-11; First posted 2024-02-07 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Sedentary Behaviour
Keywords: Sedentary behaviour; Home-office; Office work; Technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group will receive the Click2Move intervention for one year, including a wearable (provided by the research group) and mobile phone application downloaded in the participants own mobile phone. Click2Move intervention comprises elements at three levels: environmental (activity tracking and app provision, reminders, cooperative challenges, and social chat), organisational level (organisational support and motivational messages), and at individual level (educational materials, self-monitoring, feedback provision, demonstration videos and a list of strategies).
  Interventions: Behavioral: Click2Move
- Control group (No Intervention): Participants in the control arm will be asked to complete the same study measurements as those in the intervention arms, at the same time points. The control arm participants will not receive any device, nor will they have to download the mobile phone application. After the year of the intervention, they will be able to receive the intervention if they agree.

INTERVENTIONS:
Behavioral: Click2Move — One year multicomponent intervention including a wearable, and a mobile phone application downloaded in the own mobile phone. Participants will have activity tracking and app provision, sedentary reminders, cooperative challenges, organisational support and motivational messages, educational material, self-monitoring, feedback provision, demonstration videos and strategies.
  Arms: Experimental group

SUMMARY:
The goal of this clinical evaluate the effectiveness of the Ckick2Move Programme, a multicomponent digital-based intervention, to reduce sedentary behaviour among home-office workers, and the impact on employees physcial activity patterns, musculoskeletal risk and work-related outcomes (i.e., absenteeism, presenteeism, occupational fatigue and job satisfaction). The study will take place in four countries along Europe (Spain, Ireland, Netherlands, and Slovenia).

DETAILED DESCRIPTION:
This study will be conducted, analysed, and reported according to the Consolidation Standards of Reporting Trials (CONSORT) statement for cluster RCTs. A two-arm cluster randomised controlled trial will be undertaken. Participants will be randomised by cluster to receive the intervention or act as a control group and maintain their usual work. The protocol was approved by the Research Ethics Committee of the University of Vic - Central University of Catalonia (278/2023).

The primary objectives are a) to evaluate the effectiveness of the Click2Move intervention on reducing occupational sedentary time in home-office workers, and b) to assess the process evaluation of the Click2Move intervention in hybrid office workers.

The secondary objectives are a) to investigate whether the Click2Move intervention impacts on employee's physical activity and sedentary behaviours, and b) to evaluate the impact of the Click2Move intervention on employees' musculoskeletal health and work-related outcomes.

Sample size: Based on an assumed mean reduction of 55.92 minutes/day sitting in the intervention group and a standard deviation in both groups of 90 minutes/day, a power of 80%, a two-sided alpha of 0.05, and a 20% dropout rate, we need 200 participants across 4 companies at baseline. Within each company, randomization in the intervention group or control group takes place at the unit level (clusters) through a hierarchic clustering between units in a company, assuming a low intra-cluster correlation coefficient (ICC) of 0.05 for the unit and 0.2 for the company. Per company, 1 control unit and 1 intervention unit will be included with the total number of participants being equal per company (n=50). The total sample size will be equally distributed across both conditions (intervention group or control group).

Recruitment process: Each national coordinator will send a first email to potential country-representative companies from a variety of sectors in their own language with a flyer and a short survey with the eligible companies' criteria. This email will have attached the company information statement. Those who expressed their interest to participate will receive an email (if they meet the inclusion criteria) to organise an appointment to explain the project in greater detail and resolve any possible doubts or issues the company may have. If a commitment is made, the company will have access to the overall materials of the programme. As for the participants recruitment, the company will receive a template email to share with their own workers. This email will contain a flyer and a link with a short survey, including the information statement and the informed consent. The national coordinator will review all the responses and will identify those that meet the eligibility criteria. Those participants who meet the inclusion criteria and signed the informed consent digitally through the survey, will be included in a list of participants. Subsequently, they will receive a second email to thank them for their interest and will be invited to make a group appointment in the company for the baseline assessments in March (first meeting). This email will contain a link with the measurement survey participants will be asked to complete before the appointment. Those participants who have not answered the survey will be asked to answer it during the meeting.

Allocation: After baseline measurements take place (March 2024) participants will be randomised by clusters (units) 1:1, to either intervention or control group at the company level to reduce the risk of contamination. The randomisation will be taken by the principal investigator. Participants will receive information according to the allocated group the last week of March by email. Participants allocated in the intervention group, will be arranged for a second group meeting in the company on the first week of April 2024, where they will be provided with an activity tracker, the App link with the username and password accompanied by a usage tutorial. The control group will not attend a second meeting. Control group participants will not receive any device, nor will they have to download the mobile phone application. After the year of the intervention, they will be able to receive the intervention if they choose.

Blinding: Given the nature of the study, it is not possible to blind participants to which intervention they receive. However, the randomisation will be taken at the unit level to reduce the risk of contamination. Measurement team members will not be blinded to group allocation.

Intervention: The Click2Move intervention consists of a mobile phone application (C2M App) compatible with Android and iOS in combination with a wearable monitor (an activity tracker) provided by the project. Click2Move is a multicomponent intervention that covers behavioural change elements at the social environmental, organisational, and individual level.

The C2M App will be downloaded in the intervention group participants' devices. They will access the App using their email address and the password received during the second meeting (April 2024). An initial wizard will guide the user through the activity tracker synchronization. The App will include a wide range of functionalities:

* Profile page: In the profile page users will be able to change their password and edit their profile including an avatar. Initially established working hours and days could be modified through the profile page. Finally, in this section, users will have the opportunity to share any comment, suggestion, or concern about the programme to their company.
* Self-monitoring and feedback provision: Time spent in a sedentary behaviour and the number of steps will be recorded in real-time through the activity tracker during the pre-established working hours. Once users open the C2M App, data will be synchronized and displayed through the "Home" page: number of steps, sedentary time, sedentary reminders (accepted and refused) and additional strategies for breaking sedentary time that they selected as completed without receiving reminders. This information will be visualised through a loop and the actual number records. Moreover, activity and sedentary history will be visualised through the "History" page.
* Strategies: The "Strategies" section will include a list of two different types of strategies: specific and general strategies. Strategies preferred by the participants can be marked as "liked", and the most popular strategies will appear on the bottom of the different sections.

  * Specific strategies have the aim to break sitting time, requiring a minimum of movement from 1 to 5 minutes, containing different categories: walk, stretch, strength, mobility, stability or combination (i.e., including more than one of the above). Each strategy will contain an image, a tittle and description of the exercise, including the benefits of doing that exercise, the development instructions, the number of repetitions, and a video demonstration.
  * General strategies have the aim to reduce total sitting time during working or non-working hours (e.g., walking meetings).
* Sedentary reminders: Every hour without moving from the chair, participants will receive a reminder through a vibration of the activity tracker. After that, the user will have to open the App, where a message to invite him/her to break sedentary time and perform the proposed specific strategy, they will be able to accept or skip it. Employees who not receive reminders (i.e., they are sufficiently active), will receive a motivational message where users will be able to select the strategies that they have implemented during this day from those proposed or additionally select others for non-described strategies. Users will receive a push notification encouraging them to break their sitting time in case they ignored all the reminders.
* Cooperative challenges: These challenges will be done among all company workers who participate in the programme. Examples of the challenges include: to achieve a pre-determined number of steps during a month or that an individual does not receive more than a pre-determined number of inactivity reminders during a period. The duration of the challenges will not be more than a month. For each challenge, the tittle, the description of the challenge, and the duration (start date and end date) will appear. Moreover, in the challenge requirements will appear the achievement of the challenges among all the participants and the individual contribution to the challenge.
* Motivational messages: Once the challenge is completed, users will receive a motivational message (e.g., good job, you have done 6000 steps during the working day), which will be signed by the managers. Each challenge will include a forum where users will be able to share their experiences with other employees. Additionally, the company will select an individual from each department who will be the facilitator of the forum, encouraging participation in the challenges and leading by example.

In parallel to the C2M App, intervention group participants will receive email communication at two levels: a) An initiation email from the company with an encouraging video from the CEO or staff leader of a similar rank and Periodic (monthly), and b) emails send by the C2M team with educational material (videos and infographics) showing the benefits of reducing occupational sedentary behaviour.

Data collection: Data will be collected at four time points for both intervention and control group participants: at baseline (March 2024), after 3 months (June 2024), 6 months (September 2024), and 12 months (March 2025) to both groups. Self-report questionnaires will be delivered through the REDCap (Research Electronic Data Capture) via email prior to the face-to-face appointment. In this meeting, trained researchers will provide participants with the activPAL device and the diary log. The researcher will ensure that participants have completed the questionnaires online, otherwise they will be asked to complete them in the meeting.

Data management: Data will be measured by each country and collected centrally by the REDCap project platform allocated at the UVic-UCC server. Our data management plan will align with the FAIR data principle for its data management approach (Findability, Accessibility, Interoperability, and Reusability). Data management will also align with all EU General Data Protection Regulations (GDPR).

Data analysis: Data will be assessed for normality using the Kolmogorov-Smirnov method, with manual inspection of histograms and box plots for the whole group and within clusters. Descriptive characteristics for demographic, work environment, behavioural measures, health and work will be described using frequencies, mean and standard deviations and median and interquartile range. Independent samples t-tests (or the non-parametric Mann-Whitney U test) will be used to determine differences between clusters at baseline. Linear mixed models, accounting for any covariates (including baseline values), will be employed to determine the effects of the intervention. Effect sizes will be calculated by dividing the difference in group means by the average standard deviation of the pooled data. All statistical analysis will be conducted using STATA MP (StataCorp, College Station, TX, USA) or SPSS (v 28, IBM, Chicago, IL, USA). For the process evaluation, questionnaire data will be summarised using frequency counts and means (± SD) where appropriate. Audio-recordings of focus groups will be transcribed verbatim and analysed using the principles of Thematic Analysis. MAXQDA 2024 (HRB 78781, AG Berlin Charlottenburg, Germany) will be employed for the qualitative analysis.

Financial disclose: The Click2Move Project was funded by the Erasmus+ Programme call: ERASMUS-SPORT-2021-SCP, grant number 101050490.

ELIGIBILITY:
Inclusion Criteria:

* Companies inclusion criteria: a) companies' size >50 employees, b) with home-office policies, and c) having different units.
* Participants inclusion criteria: Adults, full or part-time home-office work, working from home at least 2 days per week, able to walk without the use of an assistive device or requiring assistance from another person.

Exclusion Criteria:

* Companies exclusion criteria: Involving in other initiatives to reduce sedentary behaviour.
* Participants exclusion criteria: Unable to read and understand language. Employees with an end date for employment until after the study has been completed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Occupational sitting time | Baseline, 3 months, 6 months and 12 months.
  The activPAL3TM (PAL Technologies Ltd., Glasgow, UK) will be used to measure and quantify the occupational sedentary behaviour patterns of employees. This device is a valid measure to quantify body posture and activity patterns during free-living conditions.
  Participants will wear the activPAL3TM for 7 days. Additionally, participants will be asked to record their daily wake-up time, bedtime, working hours, and any monitor removal time through a diary log.
Leisure sitting time | Baseline, 3 months, 6 months and 12 months.
  The activPAL3TM (PAL Technologies Ltd., Glasgow, UK) will be used to measure and quantify the leisure sedentary behaviour patterns of employees. This device is a valid measure to quantify body posture and activity patterns during free-living conditions.
Total sitting time | Baseline, 3 months, 6 months and 12 months.
  The activPAL3TM (PAL Technologies Ltd., Glasgow, UK) will be used to measure and quantify the leisure sedentary behaviour patterns of employees. This device is a valid measure to quantify body posture and activity patterns during free-living conditions.

SECONDARY OUTCOMES:
Occupational physical activity (MVPA, LIPA and stepping) | Baseline, 3 months, 6 months and 12 months.
  The activPAL3TM (PAL Technologies Ltd., Glasgow, UK) will be used to measure and quantify the occupational physical activity patterns of employees. This device is a valid measure to quantify body posture and activity patterns during free-living conditions.
  Participants will wear the activPAL3TM for 7 days. Additionally, participants will be asked to record their daily wake-up time, bedtime, working hours, and any monitor removal time through a diary log.
Leisure-time physical activity (MVPA, LIPA and stepping) | Baseline, 3 months, 6 months and 12 months.
  The activPAL3TM (PAL Technologies Ltd., Glasgow, UK) will be used to measure and quantify the occupational physical activity patterns of employees. This device is a valid measure to quantify body posture and activity patterns during free-living conditions.
  Participants will wear the activPAL3TM for 7 days. Additionally, participants will be asked to record their daily wake-up time, bedtime, working hours, and any monitor removal time through a diary log.
Total physical activity (MVPA, LIPA and stepping) | Baseline, 3 months, 6 months and 12 months.
  The activPAL3TM (PAL Technologies Ltd., Glasgow, UK) will be used to measure and quantify the occupational physical activity patterns of employees. This device is a valid measure to quantify body posture and activity patterns during free-living conditions.
  Participants will wear the activPAL3TM for 7 days. Additionally, participants will be asked to record their daily wake-up time, bedtime, working hours, and any monitor removal time through a diary log.
Occupational standing time | Baseline, 3 months, 6 months and 12 months.
  The activPAL3TM (PAL Technologies Ltd., Glasgow, UK) will be used to measure and quantify the occupational physical activity patterns of employees. This device is a valid measure to quantify body posture and activity patterns during free-living conditions.
  Participants will wear the activPAL3TM for 7 days. Additionally, participants will be asked to record their daily wake-up time, bedtime, working hours, and any monitor removal time through a diary log.
Leisure standing time | Baseline, 3 months, 6 months and 12 months.
  The activPAL3TM (PAL Technologies Ltd., Glasgow, UK) will be used to measure and quantify the occupational physical activity patterns of employees. This device is a valid measure to quantify body posture and activity patterns during free-living conditions.
  Participants will wear the activPAL3TM for 7 days. Additionally, participants will be asked to record their daily wake-up time, bedtime, working hours, and any monitor removal time through a diary log.
Total standing time | Baseline, 3 months, 6 months and 12 months.
  The activPAL3TM (PAL Technologies Ltd., Glasgow, UK) will be used to measure and quantify the occupational physical activity patterns of employees. This device is a valid measure to quantify body posture and activity patterns during free-living conditions.
  Participants will wear the activPAL3TM for 7 days. Additionally, participants will be asked to record their daily wake-up time, bedtime, working hours, and any monitor removal time through a diary log.
Presenteeism | Baseline, 3 months, 6 months and 12 months
  Health and Work Performance Questionnaire, which showed its validity, but also its reliability and sensitivity to change. Two questions that ask employers to rate working in their job on a 0-10 scale of work performance (worst to best), and rank themselves over the past 4 weeks during the time they were at work. Absolute presenteeism will be calculated as the difference between the score for self over the past 4 weeks and the score for the average worker in the same job. A higher score indicated lower amount of lost performance.
Occupational fatigue | Baseline, 3 months, 6 months and 12 months
  Need for Recovery scale was shown to be valid to measure occupational fatigue and showed a good psychometric quality. Additionally, the Need for Recovery scale has shown favourable test-retest reliability and sensitivity to detect change. The Need for Recovery comprises of eleven items with yes/no answering categories. A score is calculated by adding all the scores of the individual items and transforming these into a scale from 0 to 100. Higher scores indicate a higher need for recovery after work.
Job satisfaction | Baseline, 3 months, 6 months and 12 months
  Single-item 5-point Likert scale, where 1 is extremely dissatisfied and 5 extremely satisfied. The standard satisfaction scale ranging from 1 to 5 will be converted into 0 to 100 scales using the formula: AdjSS = 100 x (stsSS-1) / (5-1), where adjSS and stdSS will be "adjusted satisfaction score" and "standard satisfaction score", respectively. With the new scoring method, job satisfaction fell into 5 categories: "extremely dissatisfied" ((adjSS: 10-29), "dissatisfied" (30-49), "generally satisfied or not" (50-59), "satisfied" (70-89), and "extremely satisfied" (90-100).
Musculoskeletal symptoms | Baseline, 3 months, 6 months and 12 months
  Pain intensity will be measured through 11-point Numeric Rating Scale. Standardised Nordic Questionnaire, an internationally self-administered, will measure musculoskeletal symptoms, designed primarily in the working population, and under no circumstances was it designed for clinical diagnosis. The general questionnaire consists of 8 questions with dichotomous and Likert-type (4 to 5 levels of response) answers. The questions refer to the presence of discomfort, its duration and each episode of pain, the duration of temporary disability, the need for treatment, and the cause of discomfort. The Standard Nordic Questionnaire has proved to be valid, realiable and feasible tool that allows musculoskeletal problems among different anatomical areas in epidemiological and ergonomic studies.
Absenteeism | Baseline, 3 months, 6 months and 12 months
  Health and Work Performance Questionnaire, which showed its validity, but also its reliability and sensitivity to change. Three open questions about how many hours participants work the past 4 weeks, how many hours the employer expects employer work in the past 7 days or in a typical 7-day week and number of entire or partial days missed in the past 4 weeks for mental or physical health, for other reasons (e.g., vacations) will be used to score the absolute absenteeism (4*hours your employer expect to work - hours did employers work the past 4 weeks). Absolut absenteeism (i.e., number of missed workdays) is scored in terms of hours lost per month, a high score indicates a higher amount of absenteeism. HPQ showed its validity, but also its reliability and sensitivity to change.

OTHER OUTCOMES:
Process evaluation | 3 months, 6 months and 12 months
  Self-reported questionnaire, at 3 months, will assess usability, acceptability, perceived usefulness and satisfaction through 7-point Likert scales. At 6 and 12 months, participant's' opinions of the intervention components will be also assessed with 7-point Likert scales.
  Participants allocated to the intervention groups (and who were still taking part in 12 month follow-up) will be also offered the opportunity (via email) to take part in a focus group to examine engagement in what worked and what did not work, and suggestions to improve, along with the impeding or enhancing factors for behaviour sustainability considering the Medical Research Council guidance (MRC) (context, implementation and mechanisms of impact) (18, 19). Separate online focus groups will be conducted for each country partner with 6-10 participants per each group.
Socio demographic | Baseline
  At baseline, participants will be asked for their: age, sex, educational level, current job role, occupational sector, length of time in post in the company, working hours, how often they usually work from home, physical work environment , commute (distance from home to work, time and transport).

CONTACTS AND LOCATIONS:
Overall Officials: Judit Bort-Roig, PhD, Principal Investigator — UVic-UCC
Locations (1):
- Arthesis Group, Manlleu, Catalonia, Spain

REFERENCES:
- [Background] Edwardson CL, Yates T, Biddle SJH, Davies MJ, Dunstan DW, Esliger DW, Gray LJ, Jackson B, O'Connell SE, Waheed G, Munir F. Effectiveness of the Stand More AT (SMArT) Work intervention: cluster randomised controlled trial. BMJ. 2018 Oct 10;363:k3870. doi: 10.1136/bmj.k3870. PMID 30305278
- [Background] Cane J, O'Connor D, Michie S. Validation of the theoretical domains framework for use in behaviour change and implementation research. Implement Sci. 2012 Apr 24;7:37. doi: 10.1186/1748-5908-7-37. PMID 22530986
- [Background] Rajkumar E, Rajan AM, Daniel M, Lakshmi R, John R, George AJ, Abraham J, Varghese J. The psychological impact of quarantine due to COVID-19: A systematic review of risk, protective factors and interventions using socio-ecological model framework. Heliyon. 2022 Jun;8(6):e09765. doi: 10.1016/j.heliyon.2022.e09765. Epub 2022 Jun 19. PMID 35756104
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] Michie S, Richardson M, Johnston M, Abraham C, Francis J, Hardeman W, Eccles MP, Cane J, Wood CE. The behavior change technique taxonomy (v1) of 93 hierarchically clustered techniques: building an international consensus for the reporting of behavior change interventions. Ann Behav Med. 2013 Aug;46(1):81-95. doi: 10.1007/s12160-013-9486-6. PMID 23512568
- [Background] Huang Y, Benford S, Blake H. Digital Interventions to Reduce Sedentary Behaviors of Office Workers: Scoping Review. J Med Internet Res. 2019 Feb 7;21(2):e11079. doi: 10.2196/11079. PMID 30730294
- [Background] Kessler RC, Barber C, Beck A, Berglund P, Cleary PD, McKenas D, Pronk N, Simon G, Stang P, Ustun TB, Wang P. The World Health Organization Health and Work Performance Questionnaire (HPQ). J Occup Environ Med. 2003 Feb;45(2):156-74. doi: 10.1097/01.jom.0000052967.43131.51. PMID 12625231
- [Background] Kessler RC, Ames M, Hymel PA, Loeppke R, McKenas DK, Richling DE, Stang PE, Ustun TB. Using the World Health Organization Health and Work Performance Questionnaire (HPQ) to evaluate the indirect workplace costs of illness. J Occup Environ Med. 2004 Jun;46(6 Suppl):S23-37. doi: 10.1097/01.jom.0000126683.75201.c5. PMID 15194893
- [Background] van Veldhoven M, Broersen S. Measurement quality and validity of the "need for recovery scale". Occup Environ Med. 2003 Jun;60 Suppl 1(Suppl 1):i3-9. doi: 10.1136/oem.60.suppl_1.i3. PMID 12782740
- [Background] de Croon EM, Sluiter JK, Frings-Dresen MH. Psychometric properties of the Need for Recovery after work scale: test-retest reliability and sensitivity to detect change. Occup Environ Med. 2006 Mar;63(3):202-6. doi: 10.1136/oem.2004.018275. PMID 16497863
- [Background] Braun, V., & Clarke, V. (2006). Using thematic analysis in psychology. Qualitative research in psychology, 3(2), 77-101.
- [Background] Nagy MS. Using a single-item approach to measure facet job satisfaction. Journal of Occupational and Organizational Psychology. 2002;75(1):77-86.
- [Background] Kuorinka I, Jonsson B, Kilbom A, Vinterberg H, Biering-Sorensen F, Andersson G, Jorgensen K. Standardised Nordic questionnaires for the analysis of musculoskeletal symptoms. Appl Ergon. 1987 Sep;18(3):233-7. doi: 10.1016/0003-6870(87)90010-x. PMID 15676628
- [Background] Powell C, Carson BP, Dowd KP, Donnelly AE. Simultaneous validation of five activity monitors for use in adult populations. Scand J Med Sci Sports. 2017 Dec;27(12):1881-1892. doi: 10.1111/sms.12813. Epub 2016 Dec 1. PMID 27905148
- [Background] Wu Y, Petterson JL, Bray NW, Kimmerly DS, O'Brien MW. Validity of the activPAL monitor to measure stepping activity and activity intensity: A systematic review. Gait Posture. 2022 Sep;97:165-173. doi: 10.1016/j.gaitpost.2022.08.002. Epub 2022 Aug 6. PMID 35964334
- [Background] Dowd KP, Harrington DM, Bourke AK, Nelson J, Donnelly AE. The measurement of sedentary patterns and behaviors using the activPAL Professional physical activity monitor. Physiol Meas. 2012 Nov;33(11):1887-99. doi: 10.1088/0967-3334/33/11/1887. Epub 2012 Oct 31. PMID 23111150
- [Background] O'Brien MW, Wu Y, Petterson JL, Bray NW, Kimmerly DS. Validity of the ActivPAL monitor to distinguish postures: A systematic review. Gait Posture. 2022 May;94:107-113. doi: 10.1016/j.gaitpost.2022.03.002. Epub 2022 Mar 7. PMID 35276456
- [Background] Moore GF, Audrey S, Barker M, Bond L, Bonell C, Hardeman W, Moore L, O'Cathain A, Tinati T, Wight D, Baird J. Process evaluation of complex interventions: Medical Research Council guidance. BMJ. 2015 Mar 19;350:h1258. doi: 10.1136/bmj.h1258. PMID 25791983
- [Background] Skivington K, Matthews L, Simpson SA, Craig P, Baird J, Blazeby JM, Boyd KA, Craig N, French DP, McIntosh E, Petticrew M, Rycroft-Malone J, White M, Moore L. A new framework for developing and evaluating complex interventions: update of Medical Research Council guidance. BMJ. 2021 Sep 30;374:n2061. doi: 10.1136/bmj.n2061. PMID 34593508
- [Background] Liu JA, Wang Q, Lu ZX. Job satisfaction and its modeling among township health center employees: a quantitative study in poor rural China. BMC Health Serv Res. 2010 May 10;10:115. doi: 10.1186/1472-6963-10-115. PMID 20459725
- [Derived] Bort-Roig J, Pares-Salomon I, Loef B, Vaque-Crusellas C, Coffey A, Gustems-Morral A, Sene-Mir AM, Luznik I, Pajek M, Dowd KP, Puig-Ribera A, Proper KI. A digital intervention to reduce home-office workers' sedentary behaviour: protocol for the evaluation of the Click2Move programme, a cluster randomised controlled trial. BMC Public Health. 2025 Jan 30;25(1):387. doi: 10.1186/s12889-025-21598-7. PMID 39885479